CLINICAL TRIAL: NCT02270528
Title: Acute Effects of High Intensity Interval Exercise on Executive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM20000451
Record Dates: First submitted 2014-09-25; First posted 2014-10-21 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: High Intensity Interval Exercise (HIIE); Pain Perception; Wisconsin Card Sorting Task
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIT1 (Experimental): This group will participate in the Wisconsin Card Sorting Task (WCST) two times. During the first attempt, prior to the WCST, this group will perform a warm-up and the high intensity interval exercise. The second attempt, prior to the WCST, this group will perform a warm-up and 5-minute stationary period. All measures of independent variables (pH, lactate, RPE, RPP, and FS) will be the same for all groups.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive Task
- HIT2 (Experimental): This group will participate in the Wisconsin Card Sorting Task (WCST) two times. During the first attempt, prior to the WCST, this group will perform a warm-up and a 5-minute stationary period. The second attempt, prior to the WCST, this group will perform a warm-up and the high intensity interval exercise. All measures of independent variables (pH, lactate, RPE, RPP, and FS) will be the same for all groups.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive Task
- CON (Other): This group will participate in the Wisconsin Card Sorting Task (WCST) two times. During the first attempt and second attempt, prior to the WCST, this group will participate in a 15-minute stationary period. All measures of independent variables (pH, lactate, RPE, RPP, and FS) will be the same for all groups.
  Interventions: Behavioral: Cognitive Task

INTERVENTIONS:
Behavioral: Exercise — 10 seconds of sprinting on a bicycle ergometer against a resistance equivalent to 5.5% of a participant's body weight, followed by 20 seconds of rest, repeated 10 times. (~5 minutes)
  Arms: HIT1; HIT2
Behavioral: Cognitive Task — The Wisconsin Card Sorting Task (WCST) is a measure of Executive Function.

SUMMARY:
This study will examine the acute effects of high intensity interval ergometry on peripheral concentrations of lactate and hydrogen ions, as well as cognitive function. Approximately 60 healthy, college-aged males will participate in the Wisconsin Card Sorting Task (WCST), a measure of executive function, two times over a span of two weeks. Prior to the WCST, participants will complete either a warm-up, a warm-up and high intensity interval exercise, or a stationary period. Changes in lactate, pH, and WCST score will be evaluated between and within groups in relation to the presence of the high intensity exercise stimulus.

DETAILED DESCRIPTION:
The experimental protocol will be performed in three groups. Two of the three groups (HIT1 and HIT2) will counterbalance one another, meaning these participants will each receive the same level of treatment, but the treatments will occur in different sequence. The third group will serve as the control (CON). All qualified subjects will complete a consent form after receiving a detailed explanation of the experimental purpose and procedure by the investigator. Subjects qualify to participate in this study based upon the results of the preliminary health history record, ACSM risk assessment, and a 7-day activity recall form IPAQ. Following consent, participants will be randomized into one of three groups and will be scheduled three(3) lab sessions. A Subject Tracking Form will be used to monitor the progress of each subject.

All three groups begin the study with the same session protocol, constituting Day 1 (Baseline). This session will include baseline measurements of perceived effort (RPE), perceived pain (RPP), and affect (FS). These measures will be taken before and after the maximal oxygen uptake test scheduled on this day. Two single 15 mL blood samples (~1 tablespoon) will be drawn for baseline pH and lactate quantification. Blood draws (BD) are repeated for a total of 8 times throughout the study for a total of 120 mL of blood. During the two experimental sessions (Session 2 and Session 3) blood will be drawn 3 times each; prior to HIT or seated rest, immediately following HIT or seated rest, and following the Wisconsin Card Sorting Task (WCST). The seventh and eight blood draws will occur during baseline, immediately before and after the maximal oxygen uptake exercise test. Each group will participate in all 8 blood draws. A demonstration of the WCST and a review of the Tabata high-intensity interval training protocol (HIT) will also be given during this session. Session 1 includes a cardiovascular fitness assessment (relative VO2 test) and body fat assessment (Bioelectrical Impedence Analysis, or BIA).

The following two sessions, Day 3 (Session 2) and Day 17 (Session 3), will be different for each group. The first group, (HIT1), will complete a warm-up, HIT, and the WCST during Session 2. The next session, Session 3, will be scheduled no less than 14 days from Session 2 and includes a warm-up, a 5-minute stationary period, and the WCST. The second group, (HIT2), will complete the same protocols as HIT1, but will complete Session 2 and Session 3 in reverse order. The control group (CON) will not perform the warm-up or the HIT exercise before either WCST. This group will still have 14-days separating WCST attempts. A follow-up by email will be used to report the results of the WCST scores to each participant once all subjects have completed the study in its entirety. Instructions on how to receive compensation for participating in the study will also be provided in the follow-up.

Data will be analyzed using the current version of SPSS Statistics. A 2 (HIT, no HIT) x 3 (pre-, immediately post-, and delayed post- HIT) repeated measures ANOVA will be used to determine the affects of HIT on biophysiological functions (La, H+, RPP, RPE, and FS). A paired t-test will show changes in executive function due to HIT. A Pearson correlation will determine the influence of biophysiological factors on cognitive function and a 3 (HIT1, HIT2, CON) x 2 (time of WCST) mixed-model ANOVA will demonstrate the learning effects associated with the WCST over a 14-day period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male college students
* Ages of 18-35 years old
* Body fat percent < 25%

Exclusion Criteria:

* Moderate to high risk for cardiovascular disease
* Reporting any known physical or psychological diseases or disorders
* Participating in certain prescription and/or illegal drug use
* Smoking
* Body fat percent > 25%
* Those having undergone any surgery, serious injury, or hospitalization within the past five years
* Those having experienced a major life event (eg divorce, family death) in the past five years

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Peripheral Blood Lactate | 8 times total; 2 at Baseline (Day 1; Minute 14 and Minute 29), 3 in session 1 (Day 3; Minute 2, Minute 18, and Minute 29), and 3 in session 2 (Day 17; Minute 2, Minute 18, and Minute 29); Maximum Time Frame at Session 2 (Day 17, Minute 29)
  Lactate is known to increase during exercise. At each time frame, ~15mL of blood will be sampled from a subject via intravenous catheter. From this sample, blood will be analyzed for lactate using a YSI2300.
Peripheral Hydrogen Ions, Peripheral Blood pH | 8 times total; 2 at Baseline (Day 1; Minute 14 and Minute 29), 3 in session 1 (Day 3; Minute 2, Minute 18, and Minute 29), and 3 in session 2 (Day 17; Minute 2, Minute 18, and Minute 29); Maximum Time Frame at Session 2 (Day 17, Minute 29)
  pH decreases during rigorous or intense exercise. At each time frame, ~15mL of blood will be sampled from a subject via intravenous catheter. From this sample, blood will be analyzed for Hydrogen Ions (pH) via a pH electrode.
Executive Function | 2 times total, 1 in session 1 (Day 3; Minute 20), 1 in session 2 (Day 17, Minute 20); Maximum Time Frame at Session 2 (Day 17, Minute 20)
  Executive Function deals with the ability to problem solve, plan, and make decisions. The Wisconsin Card Sorting Task (WCST) is a computerized version of a task of executive function. Categories completed will be used as the measure of executive function ability.

SECONDARY OUTCOMES:
Ratings of Perceived Pain (RPP) | 8 times total; 2 at Baseline (Day 1; Minute 15 and Minute 30), 3 in session 1 (Day 3; Minute 3, Minute 19, and Minute 30), and 3 in session 2 (Day 17; Minute 3, Minute 19, and Minute 30); Maximum Time Frame at Session 2 (Day 17, Minute 30)
  This is a visual analog scale used to determine an individual's relative perceived level of pain. The individual will mark on the scale how much pain they are experiencing.
Ratings of Perceived Exertion (RPE) | 8 times total; 2 at Baseline (Day 1; Minute 15 and Minute 30), 3 in session 1 (Day 3; Minute 3, Minute 19, and Minute 30), and 3 in session 2 (Day 17; Minute 3, Minute 19, and Minute 30); Maximum Time Frame at Session 2 (Day 17, Minute 30)
  RPE will be measured using Borg's scale of exertion. This is a numeric scale (6-20). An individual will state the number that correlates to the level of effort being given.
Emotion (Feeling Scale, FS) | 8 times total; 2 at Baseline (Day 1; Minute 15 and Minute 30), 3 in session 1 (Day 3; Minute 3, Minute 19, and Minute 30), and 3 in session 2 (Day 17; Minute 3, Minute 19, and Minute 30); Maximum Time Frame at Session 2 (Day 17, Minute 30)
  This is a numeric scale (-5 to +5). An individual will state the number that correlates to the emotion being felt (-5= Very Bad to +5+Very Good).

CONTACTS AND LOCATIONS:
Overall Officials: Edmund O Acevedo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Clinical Research Unit, MCVH-VCU, Richmond, Virginia, United States